CLINICAL TRIAL: NCT02173028
Title: RESynchronizaTiOn theRapy and bEta-blocker Titration : RESTORE
Brief Title: RESynchronizaTiOn theRapy and bEta-blocker Titration
Acronym: RESTORE
Status: Completed | Type: Observational
Sponsor: Giuseppe Ricciardi (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Ricciardi, Principal Investigator, University of Florence
Organization: University of Florence (Other)
Other Study IDs: Rif. n. 89/11 - 2011/0043537
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Beta Blocker Intolerance; Congestive Heart Failure
Keywords: Beta Blocker Intolerance;; Remote Patient Management system;; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Optimal beta blocker titration: We will compare the efficacy of two management strategies for beta-blocker up-titration: Standard in-office visits vs. Remote follow-up.
- Without optimal titration of beta blocker: This analysis will be conducted within the Cardiac Resynchronization Therapy observational study Modular Registry (CRT MORE - ClinicalTrials.gov Identifier: NCT01573091).

SUMMARY:
Patients will be treated according to the clinical practice of the participating centers and to the international guidelines for the treatment of heart failure.The present analysis provides a collection of data about the changes to drug therapy after the "Cardiac Resynchronization Therapy" (CRT) procedure , and any signs and symptoms of intolerance to prescribed medications.

DETAILED DESCRIPTION:
The treatment of chronic heart failure is currently based on the use of ACE (Angiotensin Converting Enzyme) inhibitors and beta-blockers. Although this therapy is universally accepted up to 10-20% of patients may be intolerant. Moreover, the majority of patients are not treated with the doses that have been shown to be effective in controlled clinical trials. Although it is possible that even low doses of neurohumoral inhibitors are still effective than placebo, a greater benefit can be obtained at maximum doses. Therefore, it is generally recommended that these agents are used at recommended doses found to be effective in controlled studies. There are many reasons for the lack of prescription neurohumoral inhibitors and their use in non-optimal doses. These include both an inadequate clinical management, and low tolerance to drugs. As far as beta-blockers, their poor tolerability has at least two main causes: 1) the effects not related to heart failure (eg, bradycardia, AtrioVentricular (AV) block, bronchial asthma), 2) the acute negative inotropic effects, which can cause a further deterioration of hemodynamic parameters.

The primary objective of the analysis is to demonstrate that cardiac resynchronization therapy (CRT) may allow titration of beta-blockers (carvedilol or bisoprolol) until the optimal dosage, or at least to the effective dose, in patients with heart failure treated to maximal doses of beta-blockers and with the indications for CRT according to current international guidelines.

The secondary objective is to evaluate the effectiveness of remote monitoring with a telemedicine system to facilitate the automatic titration of beta-blockers in comparison with the standard approach, which consists of periodic outpatient visits. The strategy adopted will depend on the availability of remote monitoring systems and standard clinical practice of each participating center.

In addition, we will evaluate the clinical response to CRT, depending on the optimal or sub-optimal dosage of beta-blockers.

ELIGIBILITY:
Inclusion Criteria:

* Patients on optimal therapy for heart failure (diuretics, ACE inhibitors and aldosterone antagonists), with stable dose in the previous month;
* Successfully implanted with CRT-D according to current European Society of Cardiology (ESC) guidelines;
* New York Heart Association (NYHA) functional class: II, III and IV;
* Left Ventricular Ejection Fraction (LVEF) ≤ 35%;
* Duration of ventricular depolarization wave (QRS) ≥ 120ms (NYHA III or IV) or ≥ 150ms in NYHA II;
* Patients with chronic atrial fibrillation will be eligible for the study only if they undergo ablation ;
* 18 years or above

Exclusion Criteria:

* Failure to comply with the scheduled follow-up;
* Life expectancy less than 12 months ;
* Pregnant women;
* Tricuspid valve mechanics;
* Severe aortic stenosis or other valve disease ;
* Patients already receiving CRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients successfully implanted with CRT-D according to current European guidelines, on optimal therapy for heart failure (diuretics, ACE inhibitors and aldosterone antagonists), with stable dose in the previous month.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Optimal beta-blockers titration due to CRT | 3 months
  The primary objective of the analysis is to demonstrate that cardiac resynchronization therapy (CRT) may allow titration of beta-blockers (carvedilol or bisoprolol) until the optimal dosage, or at least to the effective dose, in patients with heart failure treated to maximal doses of beta-blockers and with the indications for CRT according to current international guidelines.The goal is to achieve the optimal dosage of 10mg/die of bisoprolol or 50mg/die of carvedilol, or at least the recommended dose (carvedilol 37.5 mg / day or bisoprolol 7.5 mg), as shown in international treatment guidelines.

SECONDARY OUTCOMES:
Beta-blocker Titration with telemedicine system | 3 months
  The secondary objective is to evaluate the effectiveness of a Remote Patient Management (RPM) system to optimize the titration of beta-blockers in comparison with the standard approach, which consists of periodic in -hospital visits.
Clinical response to CRT | 12 months
  The response will be measured at 3 and 12 months in terms of:
  1. Amount of reverse remodeling of the left ventricle;
  2. Changes in NYHA (New York Heart Association) functional class;
  3. Ventricular arrhythmias treated by the Implantable Cardioverter Defibrillator (ICD);
  4. Adverse cardiovascular events (cardiovascular hospitalization, heart failure hospitalization) and mortality from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Gronda, Principal Investigator — MultiMedica
Locations (4):
- Italy (4):
  - Policlinico Casilino, Rome, RM
  - Ospedale Monaldi SUN, Napoli
  - Ospedale Monaldi, Napoli
  - Policlinico Federico II, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Onofrio A, Palmisano P, Rapacciuolo A, Ammendola E, Calo L, Ruocco A, Bianchi V, Maresca F, Del Giorno G, Martino A, Mauro C, Campari M, Valsecchi S, Accogli M. Effectiveness of a management program for outpatient clinic or remote titration of beta-blockers in CRT patients: The RESTORE study. Int J Cardiol. 2017 Jun 1;236:290-295. doi: 10.1016/j.ijcard.2017.02.015. Epub 2017 Feb 5. PMID 28188000